CLINICAL TRIAL: NCT06698120
Title: Assessment of Efficacy and Safety of Awake Prone Positioning in Sickle Cell Anemia Patient Admitted in Intensive Care Unit for Severe Acute Chest Syndrome
Brief Title: Awake Prone Positioning for Severe Acute Chest Syndrome
Acronym: PRONE-ACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP231628; 2023-A02167-38 (Other: IDRCB ANSM)
Record Dates: First submitted 2024-04-24; First posted 2024-11-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Chest Syndrome; Sickle Cell Anemia
Keywords: Acute Chest Syndrome; Sickle Cell Anemia; Awake Prone Positioning; Electric Impedance
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Awake prone positioning (Experimental)
  Interventions: Procedure: Awake prone positioning (APP)

INTERVENTIONS:
Procedure: Awake prone positioning (APP) — * APP are realized following the diagnosis of ACS
  * Prone positioning or supine positioning are performed under supervision of a physician or a nurse
  * Maximum session duration: 16 hours per day
  * Sessions of prone positioning can be shortened, if necessary (30 minutes minimum), for better tolerance
  * Tolerance of prone positioning is assessed by the physician in charge and sessions and may be stopped in case of poor tolerance

SUMMARY:
Acute chest syndrome (ACS) is the leading cause of admission to intensive care and the leading cause of death in patients with sickle cell disease. Irrespective of the cause of ACS, there is an heterogeneity in pulmonary ventilation/perfusion ratios, leading to worsening of the disease.

Efficiency of awake prone positioning (APP) in acute respiratory failure (ARF) was particularly highlighted during the COVID-19 pandemic. Several physiological factors contribute to this benefit including an improvement in ventilatory drive and gas exchange.

The investigator hypothesize that APP could lead to clinical improvement in ACS in terms of oxygenation and ventilatory drive, by improving the heterogeneity of ventilation

DETAILED DESCRIPTION:
* Several physiological mechanisms contribute to the benefit of APP during ARF. In addition to hypoxemia improvement, there is also an effect on ventilatory drive, notably in terms of polypnea, ROX index and inspiratory effort.
* Considering that hypoxemia in ACS contributes to the physiopathological process: deoxygenation of haemoglobin S - red blood cells falciformisation - vaso-occlusive event, APP could be an additional therapy in severe ACS. In addition, improving ventilation-perfusion ratios, mainly by recruiting dorsal zones, could be particularly useful in ACS, where pulmonary damage predominates in gravito-dependent zones.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Major sickle cell anemia (SS, SC, Sβ)
* Admission in intensive care unit for ACS
* Registered in the French social insurance regime.
* Written, informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Immediate need for intubation
* Impaired vigilance status (Glasgow scale score < 12)
* Pneumothorax
* Haemodynamically unstable
* Thoracic trauma admission
* Severely obese with body-mass index higher than 40 kg/m²
* EIT contraindication: pacemaker, automatic implantable defibrillators, skin lesions facing the EIT belt, unstable rachis fracture or medullary lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The total duration of APP during the stay in intensive care unit | 28 days

SECONDARY OUTCOMES:
Changes in respiratory parameters | Up to 28 days
  Assessment of respiratory parameters changes
GI measured by EIT | Up to 28 days
ΔEELI measured by EIT | Up to 28 days
Pain measurement assessed by visual analog scale, | Up to 28 days
Pain measurement assessed by morphine consumption | Up to 28 days
Pain measurement assessed by analgesic therapeutic escalation | Up to 28 days
Occurrence of skin lesions during the intensive care unit stay | 28 Days
Occurrence of displacement of devices during the intensive care unit stay | 28 Days
Occurrence of use of vital support therapy during the intensive care unit stay | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Turpin, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Muriel Fartoukh, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Alexandre Elabbadi, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Intensive Réanimation TENON, Paris, France

IPD SHARING:
Plan to Share IPD: No